CLINICAL TRIAL: NCT03025256
Title: Phase I/Ib Study of Concurrent Intravenous and Intrathecal Nivolumab for Melanoma and Lung Cancer Patients With Leptomeningeal Disease (LMD)
Brief Title: Intravenous and Intrathecal Nivolumab in Treating Patients With Leptomeningeal Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0567; NCI-2018-01211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0567 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acral Lentiginous Melanoma; Central Nervous System Melanoma; Clinical Stage IV Cutaneous Melanoma AJCC v8; Leptomeningeal Neoplasm; Melanocytoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Melanoma; Metastatic Mucosal Melanoma; Metastatic Uveal Melanoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Meningeal Neoplasms; Nevus; Carcinoma, Non-Small-Cell Lung; Melanoma; Uveal Melanoma; Lung Neoplasms | interventions — Specimen Handling; Spinal Puncture; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IT over 5 minutes on day 1 of every cycle. Beginning in cycle 2, patients also receive nivolumab IV over 30 minutes on day 1 (4 hours after the IT dose). Cycles repeat every 14 days for 18 cycles and then every 28 days (cycles 19 and beyond) in the absence of disease progression or unacceptable toxicity. Patients will have CSF and blood specimen collection on days 1, 2, 8 of each cycle and end of treatment. Patients undergo CT or PET at baseline, cycle 5 and then every 8 weeks. Patients undergo MRI at baseline, cycles 3, 5, and then every 8 weeks.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Lumbar Puncture — Undergo lumbar puncture for cerebrospinal fluid collection
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI of brain and spine
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Nivolumab — Given IV or IT
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of intrathecal nivolumab, and how well it works in combination with intravenous nivolumab in treating patients with leptomeningeal disease. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and/or recommended dose of intrathecal (IT) nivolumab in combination with systemic nivolumab treatment in melanoma and lung cancer with leptomeningeal disease (LMD).

SECONDARY OBJECTIVE:

I. To assess overall survival with combined intrathecal and systemic administration of nivolumab in this patient population.

EXPLORATORY OBJECTIVES:

I. Compare the immunological effects of this treatment on immune cells in the cerebrospinal fluid (CSF) to those observed in the peripheral blood and in non-LMD tumors.

II. Evaluation of predictors (clinical, molecular, and/or immune) of the efficacy and safety of this regimen.

III. To assess the effect of nivolumab on subsequent treatment. IV. To compare levels of nivolumab in the CSF and peripheral blood.

OUTLINE: This is a phase I, dose-escalation study followed by a phase Ib study.

Patients receive nivolumab IT over 5 minutes on day 1 of every cycle. Beginning in cycle 2, patients also receive nivolumab intravenously (IV) over 30 minutes on day 1 (4 hours after the IT dose). Cycles repeat every 14 days for 18 cycles and then every 28 days (cycles 19 and beyond) in the absence of disease progression or unacceptable toxicity. Patients will have CSF and blood specimen collection on days 1, 2, 8 of each cycle and end of treatment. Patients undergo computed tomography (CT) or positron emission tomography (PET) at baseline, cycle 5 and then every 8 weeks. Patients undergo magnetic resonance imaging (MRI) at baseline, cycles 3, 5, and then every 8 weeks.

After completion of study treatment, patients are followed up within 4 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiographic and/or CSF cytological evidence of LMD. For patient with melanoma: Must have a confirmed diagnosis of primary central nervous system (CNS) melanoma, melanocytomas or metastatic melanoma (cutaneous, acral-lentiginous, uveal and mucosal in origin), based on histological analysis of metastatic tissue and/or cancer cells, archival tissue permitted. For patients with lung cancer: non-small cell, based on histological analysis of metastatic tissue and/or cancer cells, archival tissue permitted
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of =< 2
* Patients may receive steroids to control symptoms related to CNS involvement, but the dose must be =< 4 mg per 24 hours of dexamethasone (or the equivalent). Physiologic replacement doses for adrenal insufficiency is allowed on this protocol
* Patients who have received radiation to brain and/or spine, including whole brain radiation, stereotactic radiosurgery, or stereotactic body radiation therapy (SBRT), are eligible, but must have completed radiation treatment at least 7 days prior to the start of treatment
* Patients who have been treated with an approved targeted therapy (BRAF inhibitor and/or MEK inhibitor) will be allowed to remain on concurrent approved targeted therapy. No other concomitant intrathecal therapy with another agent will be allowed. For patients that have received other systemic therapies, the minimum wash out period is as follows:

  * Patients that received previous IT therapy must have received their last treatment >= 7 days prior to the start of treatment
  * Patients who have received systemic chemotherapy must have received their last treatment >= 14 days prior to the start of treatment
  * Patients who have received an approved systemic biologic therapy (e.g. anti-PD-1, anti-CTLA4, IL2, interferon) must have received their last treatment >= 2 weeks prior to the start of treatment
  * Patients who have received any other investigational agents must have received their last treatment >= 14 days prior to the start of treatment
* For patients with lung cancer:

  * For chemotherapy: patients do not require a washout period, and can continue with chemotherapy during treatment with IT/IV nivolumab
  * Patients who have received an approved systemic biologic therapy (e.g. anti-PD-1, anti-CTLA4, IL2, interferon) must have received their last treatment >= 2 weeks prior to the start of treatment
  * Patients who have received any other investigational agents must have received their last treatment >= 14 days prior to the start of treatment
  * No other concomitant intrathecal therapy with another agent will be allowed
  * Patients who are receiving treatment to tyrosine kinase inhibitors or other targeted therapy agents do not require a washout period, and can continue with tyrosine kinase inhibitors or other targeted therapy agents during treatment with IT/IV nivolumab
* Age >= 18 years
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Absolute neutrophil count (ANC) >= 1.5 X 10^9/L
* Hemoglobin >= 9.0 g/dL
* Platelets >= 75 X 10^9/L
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5 X upper limit of normal (ULN)
* Total bilirubin: =< 1.5 X ULN (isolated bilirubin > 1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 X ULN
* Albumin >= 2.5 g/dL
* Creatinine OR =< 2 x ULN; calculated creatinine clearance OR >= 50 mL/min; 24-hour urine creatinine clearance >= 50 mL/min
* Absence of contraindication for Ommaya reservoir
* Women are eligible to participate if:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]
  * A Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40mIU/mL to confirm menopause
  * Females treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgment in checking serum FSH levels. If the serum FSH level is >40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal:

    * 1 week minimum for vaginal hormonal products (rings, creams, gels)
    * 4 week minimum for transdermal products
    * 8 week minimum for oral products
    * Other parenteral products may require washout periods as long as 6 months
  * A Women of childbearing potential agrees to use method(s) of contraception. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. Women of childbearing potential (WOCBP) must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab is up to 25 days. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product
  * Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year The investigator shall review contraception methods and the time period that contraception must be followed. Men who are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab is up to 25 days. Therefore, men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile and azoospermic men do not require contraception

Exclusion Criteria:

* Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 4 mg daily dexamethasone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Tocilizumab and vedolizumab are permitted, as are inhaled or topical steroids and adrenal replacement doses in the absence of active autoimmune disease

  * Subjects that require premedication with corticosteroids for a contrast allergy are excluded from this restriction and can proceed with enrollment
* Patients who have previously received alpha-PD-1 and/or anti-CTLA-4 will be eligible, unless they have ongoing > grade 2 adverse event (AE) side effects of such therapy. Ongoing physiologic replacement doses for adrenal and thyroid insufficiency are allowed on protocol
* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug (concurrent treatment with approved targeted therapies is allowed.)
* Pregnant or lactating female
* Subjects with major medical, neurologic or psychiatric condition who are judged as unable to fully comply with study therapy or assessments should not be enrolled
* Patients with a history of pneumonitis
* Evidence of active infections =< 7 days prior to initiation of study drug therapy (does not apply to viral infections that are presumed to be associated with the underlying tumor type required for study entry)
* Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 12 weeks prior to study drug
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) even if fully immunocompetent on antiretroviral therapy (ART)-due to the unknown effects of HIV on the immune response to combined nivolumab or the unique toxicity spectrum of these drugs in patients with HIV
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  Safety and tolerability of treatment will be assessed by vital signs, laboratory assessments, adverse events, and serious adverse events for the safety population. Adverse events will be graded by the Common Terminology Criteria for Adverse Events version 4.0. Categorical measures will be summarized using frequencies and percentages while continuous variables will be summarized using mean, standard deviation, median, minimum, and maximum.
Recommended dose of combined intrathecal (IT) and intravenous (IV) nivolumab defined as the highest dose for which the posterior probability of toxicity is closest to 30% (dose escalation part) | Up to 28 days
  The Bayesian modified toxicity probability interval method will be used to find the recommended dose.
Overall survival (OS) in patients treated with IT and IV nivolumab (dose expansion part) | Up to 2 years

SECONDARY OUTCOMES:
OS | Up to 2 years
  The Kaplan-Meier method will be used to estimate the distribution of OS from the start of study treatment, and Cox proportional hazard regression will be used to assess the relationship between OS and various covariates of interest, including but not limited to patient demographics, tumor characteristics, disease characteristics, and the expression of biomarkers.
Immunological effects of nivolumab | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabella C Glitza, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Glitza Oliva IC, Ferguson SD, Bassett R Jr, Foster AP, John I, Hennegan TD, Rohlfs M, Richard J, Iqbal M, Dett T, Lacey C, Jackson N, Rodgers T, Phillips S, Duncan S, Haydu L, Lin R, Amaria RN, Wong MK, Diab A, Yee C, Patel SP, McQuade JL, Fischer GM, McCutcheon IE, O'Brien BJ, Tummala S, Debnam M, Guha-Thakurta N, Wargo JA, Carapeto FCL, Hudgens CW, Huse JT, Tetzlaff MT, Burton EM, Tawbi HA, Davies MA. Concurrent intrathecal and intravenous nivolumab in leptomeningeal disease: phase 1 trial interim results. Nat Med. 2023 Apr;29(4):898-905. doi: 10.1038/s41591-022-02170-x. Epub 2023 Mar 30. PMID 36997799
- See also: M D Anderson Cancer Center — http://www.mdanderson.org